CLINICAL TRIAL: NCT01644838
Title: Principal Investigator
Brief Title: Effect of Hyoscine and Promethazine on Labor Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Samira Ebrahimzadeh Zagami, School of Nursing & Midwifery, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Hyoscine & Promethazin
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Labor Pain
Keywords: Hyoscine,; Promethazine,; The first stage of labor,; Labor pain
MeSH Terms: conditions — Labor Pain | interventions — Scopolamine; Promethazine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Promethazine (Experimental): 25 mg of promethazine
  Interventions: Drug: Promethazine
- Hyoscine (Experimental): 20 mg of hyoscine
  Interventions: Drug: Hyoscine

INTERVENTIONS:
Drug: Hyoscine — The samples were randomly allocated to inject of 20 mg of hyoscineIM in dilatation 3-5cm.
  Arms: Hyoscine
Drug: Promethazine — The samples were randomly allocated to inject of 25 mg of promethazine IM in dilatation 3-5cm.
  Arms: Promethazine

SUMMARY:
It is always considered to shorten the duration of delivery without compromising the mother and fetus by obstetrics. Hyoscine and Promethazine are used widely in hospital and research is very limited, with conflicting results regarding the efficacy of these two drugs. So the investigators decided to compare of effect of hyoscine N-butyl bromide and Promethazine on length of active phase of the first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 yrs,
* primiparous,
* having single fetus with cephalic presentation, gestational age 37-42 weeks,
* having no medical diseases,
* having no history of hospitalization due to psychological diseases,
* having no addiction to cigarette,
* having no complications during pregnancy such as hypertension,
* BMI< 26

Exclusion Criteria:

* bleeding
* CPD
* use of PG or Oxytocin
* fetus distress

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Effect of Hyoscine and Promethazine on labor pain | up to 9 months